CLINICAL TRIAL: NCT04542330
Title: Using BCG Vaccine to Enhance Non-specific Protection of Senior Citizens During the COVID-19 Pandemic. A Randomized Clinical Trial.
Brief Title: Using BCG to Protect Senior Citizens During the COVID-19 Pandemic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Odense Patient Data Explorative Network (Other); Odense University Hospital (Other); Municipality of Odense (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BCG-DENMARK-SENIOR
Record Dates: First submitted 2020-09-07; First posted 2020-09-09 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-03

CONDITIONS: Covid19; Non-specific Effects of Vaccines; Heterologous Immunity; Morbidity; Immunosenescence; Vaccine Preventable Disease
MeSH Terms: conditions — COVID-19; Vaccine-Preventable Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Placebo-controlled randomized trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to treatment. The physicians administering the BCG vaccine or placebo will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG-Denmark (Active Comparator): Participants that are randomized to the active comparator arm will receive an adult 0.1 ml dose of BCG vaccine (BCG-Denmark, AJ Vaccines) in the skin covering the left upper deltoid muscle.
  Each 0.1 ml dose of vaccine contains between 200,000 to 800,000 colony forming units of the live attenuated strain of Mycobacterium bovis (BCG), Danish strain 1331.
  Interventions: Biological: BCG-Denmark
- Control (Placebo Comparator): Participants randomized to the control group will receive one 0.1 ml dose sterile 0.9 % NaCl by intradermal injection in the left deltoid region.
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: BCG-Denmark — Mycobacterium bovis BCG live attenuated BCG-Denmark vaccine (AJ Vaccines, Copenhagen, Denmark) administered by intradermal injection in the left deltoid region.
  Other Names: BCG-1331; BCG-AJ; BCG-SSI
  Arms: BCG-Denmark
Biological: Saline — Participants randomized to the control group will receive one 0.1 ml dose sterile 0.9 % NaCl by intradermal injection in the left deltoid region.
  Other Names: NaCl
  Arms: Control

SUMMARY:
Background: The virus SARS-CoV-2 has spread rapidly throughout the world. Seniors are at high risk of severe COVID-19 when infected. Bacille Calmette-Guérin (BCG) is a vaccine against tuberculosis, with protective non-specific effects against other infections; significant reductions in morbidity and mortality have been reported, and a plausible immunological mechanism has been identified: "trained innate immunity". The investigators hypothesize that BCG vaccination can reduce the risk of COVID-19 and other infections among senior citizens during the COVID-19 pandemic.

Objectives: Primary objective: To reduce senior citizens' risk of acute infection during the COVID-19 pandemic. Secondary objectives: To reduce senior citizens' risk of SARS-CoV-2 infection during the COVID-19 pandemic. To reduce senior citizens' risk of self-reported respiratory illness during the COVID-19 pandemic.

Study design: A placebo-controlled randomized trial. Study population: 1900 seniors 65 years of age or above. Intervention: Participants will be randomized 1:1 to intradermal administration of a standard dose of BCG vaccine or placebo (saline).

Outcomes: Primary outcome: "Acute infection" identified either by a doctor, antibiotics use, hospitalization, or death due to infection. Secondary outcomes: Verified SARS-CoV-2 infection and self-reported respiratory illness.

With an expected incidence of "acute infection" of 20%, the trial can show a 25% risk reduction in the the intervention group versus the placebo group by including a total of 1900 individuals, 950 individuals in each group.

Risk for participants and impact: Based on previous experience and randomized controlled trials in adult and elderly individuals, the risks of BCG vaccination are considered low. If BCG can reduce the risk of acute infection in seniors by 25% it has tremendous public health importance, both during the COVID-19 pandemic and overall.

DETAILED DESCRIPTION:
INTRODUCTION One of the most recognized consequences of aging is a decline in immune function, so-called "immunosenescence". Vaccination is the most effective prophylactic intervention for infectious diseases, but due to immunosenescence, the efficacy of vaccines decreases with increasing age.

Due to immunosenescence, severe infections are more common in the elderly. Not least during the COVID-19 pandemic, it has become clear that elderly people are particularly susceptible to severe COVID-19. Strategies to strengthen senior citizens' immune system are urgently warranted.

Bacillus Calmette-Guérin (BCG) was developed as a childhood vaccine against tuberculosis, but our group has shown that it can protect against death from other infections, i.e. it has what the investigators have called non-specific effects (NSEs). In clinical studies, BCG vaccination was associated with decreased child mortality, mainly as a result of reduced neonatal sepsis and respiratory infections. In a meta-analysis commissioned by the World Health Organization (WHO), BCG was associated with a 42% (95%CI: 24-55%) reduction in child mortality.

NSEs of BCG are not limited to children. An Indonesian trial with 34 subjects aged 60-75 years reported that compared with placebo, consecutive BCG vaccination for 3 months reduced the incidence of acute upper respiratory tract infections by 80% (95% confidence interval (CI)=22-95%). In a very recent clinical trial in Greece, BCG vs. placebo to senior citizens at discharge from the hospital was associated with a significant decrease in time to first infection (p: 0.035). The incidence of new infections was 42.3% (99% CIs 31.9 53.4%) in the placebo group and 25.0% (95% CIs (16.4-36.16%) in the BCG group; most of the protection was against respiratory tract infections (odds ratio 0.20; p: 0.001). No difference in the frequency of adverse effects was found between groups. These data show that BCG vaccination is safe and can protect the elderly against infections.

Immunological studies have now provided an explanation for the observed NSEs of BCG: BCG induces epigenetic and metabolic reprogramming of innate immune cells such as myeloid cells and Natural Killer cells, leading to an increased antimicrobial activity, a process termed 'trained immunity'.

In a pilot study the investigators recently investigated whether BCG could induce innate immune training in seniors above 50 years of age in Guinea-Bissau. Two months after vaccination, BCG recipients had increased release of the pro-inflammatory innate cytokines interleukin (IL)-1β, IL-6 and TNF-α to non-specific stimuli. These effects were more pronounced among those with a positive Quantiferon test at baseline. Thus, BCG vaccination can induce a 'trained immunity' phenotype in older adults. including previously Mycobacterium tuberculosis exposed individuals.

Currently, numerous clinical trials are investigating the effect of BCG as a prophylactic treatment for health care workers of all ages. No results of these trials are available yet, but ecological analyses have suggested that countries with a functioning BCG vaccination program have lower COVID-19 mortality. Furthermore, in a very recent follow-up study of three cohorts of healthy volunteers who either received BCG in the last five years or not, BCG vaccination was safe and not associated with increased incidence of symptoms during the COVID-19 outbreak in the Netherlands. In fact, BCG vaccination was associated with a decrease in the incidence of sickness during the COVID-19 pandemic (adjusted odds ratio 0.58, P < 0.05).

The investigators hypothesize that BCG vaccination may strengthen the immune system of the senior citizens and may (partially) protect against getting infected and/or experiencing severe morbidity due to infections with SARS-CoV-2 and other infectious pathogens.

OBJECTIVES Primary objective: To reduce senior citizens' risk of acute infection during the COVID-19 pandemic. Secondary objectives: To reduce senior citizens' risk of SARS-CoV-2 infection during the COVID-19 pandemic. To reduce senior citizens' risk of self-reported respiratory illness during the COVID-19 pandemic.

HYPOTHESIS BCG vaccination of seniors will reduce the risk of acute infection by 25% over a period of 12 months.

PROJECT GROUP Christine Stabell Benn (MD, DMSc), Peter Aaby (DMSc), Anne Marie Rosendahl Madsen (MD, PhD student), Mette Bliddal (PhD), Sebastian Nielsen (MSc, statistician), and Frederik Schaltz-Buchholzer (MD, PhD), all from University of Southern Denmark. Lene Annette Norberg (MD, PhD) and Anne Grete Pilgaard from Municipality of Odense. Mihai Netea (MD, DMSc), Radboud Medical Centre, Nijmegen, The Netherlands. Tyra Grove Krause (MD, PhD), Statens Serum Institut.

METHODS Study design and follow-up A randomized placebo-controlled clinical trial. Participants will be followed for 12 months post-randomization with respect to illness, medical contacts, use of antibiotics, hospitalization and death. The follow-up will take place both through self-reporting, and through the Danish National Registers. Information on hospitalizations for infections and other medical conditions will be obtained through Denmark's National Patient Register and information on use of antibiotics from the Danish Prescription Register. Vaccination history will be acquired from the Danish Vaccination Registry at Statens Serum Institut. Furthermore, data on testing for SARS-CoV-2 and results will be obtained via the local department of clinical microbiology.

Since the Investigational Medicinal Product (IMP), the BCG vaccine, is used in this study on another indication than the one it has been approved for, this is classified as a phase III study.

Participants will be randomized 1:1 to receiving an intradermal BCG vaccine or placebo. Participants who are randomized in the active arm will receive a BCG vaccine (BCG-Denmark, AJ Vaccines, http://www.produktresume.dk/AppBuilder/login.html). The BCG vaccines will be handled in full compliance with the requirements of the Summary of Product Characteristics (SPC). Placebo will be 0.1 ml sterile 0.9 % NaCl, which has a similar color as the resuspended BCG vaccine.

All participants will receive one injection at inclusion. No further treatment of study participants will take place. BCG will be administered in the upper arm, intradermally, 0.1 ml of the suspended vaccine. Placebo will be administered in the upper arm, intradermally, 0.1 ml of sterile 0.9 % NaCl solution.

STUDY PROCEDURES The trial will be presented at information meetings and in relevant media, local newspapers and homepages and newsletters of the activity houses.

Citizens wishing to participate will be given written information and will be booked for an interview.

Day of inclusion (day 0) Study physicians, who are trained in good clinical practice and in providing intradermal vaccines, will be responsible for the inclusion of study participants. Informed consent will be obtained from all participants. Background information on participants will be collected in an electronic case report form system (REDCap). A blood sample of 5 ml will be drawn for subsequent testing for SARS-CoV-2 antibodies.

Randomization and blinding The study will be individually randomized, and placebo controlled. Randomization will be done using the REDCap tool with stratification per sex and age groups (65-74/75+ years of age) in randomly selected block sizes of 4 and 6.

The participant will be blinded to the treatment.

Day of inclusion till end of trial A short electronic questionnaire regarding health, symptoms and potential side effects will be sent to the participants biweekly.

End of trial Participants are asked to fill in a final questionnaire. A blood sample of 5 ml will be drawn for subsequent testing for SARS-CoV-2 antibodies.

The end of the trial is defined as whichever comes latest: The last participants last registration in the online data collection, or 365 days. When the study is ended, all participants receive an email with information about the intervention that they have received (BCG/placebo).

STATISTICAL ANALYSIS The primary endpoint "acute infection" will be analyzed as a recurrent time-to-event using an Andersen-Gill Cox proportional hazards regression model with time since inclusion as underlying time scale. Analyses will be done stratified by the block randomization variables sex and age group.

The secondary endpoint self-reported respiratory illness will be analyzed the same way as the primary endpoint. The other secondary outcome verified SARS-CoV-2 infection will be analyzed in a standard Cox proportional hazards model, but otherwise as described above.

When applicable (i.e. in the event that one or more participants have died during the follow-up period) a competing events analysis will be performed in addition (Fine-Gray model).

SAMPLE SIZE CALCULATION With an expected incidence of "acute infection" of 20% the trial can show a 25% reduction in the risk of acute infection in the intervention group versus the placebo group by including a total of 1890 individuals, 945 individuals in each group.

ELIGIBILITY:
Inclusion Criteria:

• In order to be eligible to participate in this study, a subject must meet the following criteria: ≥65 years old.

Exclusion Criteria:

* Known allergy to (components of) the BCG vaccine or serious adverse events in relation to prior BCG administration
* Previous Mycobacterium tuberculosis (M. tuberculosis) infection or known active or latent infection with M. tuberculosis or other mycobacterial species
* Previous confirmed COVID-19 infection
* Fever (>38 C) within the past 24 hours or suspicion of active viral or bacterial infection
* Vaccination with other live attenuated vaccine within the last 4 weeks
* Severely immunocompromised subjects. This exclusion category comprises:
* Subjects with known infection with the human immunodeficiency virus (HIV)
* Subjects with solid organ transplantation or bone marrow transplantation
* Subjects under chemotherapy
* Subjects with primary immunodeficiency
* Treatment with any anti-cytokine therapy within the last year
* Treatment with oral or intravenous steroids defined as daily doses of 10 mg prednisone or equivalent for longer than 3 months
* Active solid or non-solid malignancy or lymphoma within the prior two years
* Subjects who do not have access to e-Boks.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1700 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Rosendahl Madsen, MD, Principal Investigator — Bandim Health Project, Department of Clinical Research, Uni. Southern Denmark; Christine Stabell Benn, DMSc, Study Chair — Bandim Health Project, Department of Clinical Research, Uni. Southern Denmark
Locations (1):
- Seniorhuset, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable individual data can be shared on the basis of a data sharing proposal sent to cbenn@health.sdu.dk
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: When follow-up has been completed and the dataset have been closed
Access Criteria: Per justified request on email (cbenn@health.sdu.dk)

REFERENCES:
- [Background] Benn CS, Fisker AB, Rieckmann A, Sorup S, Aaby P. Vaccinology: time to change the paradigm? Lancet Infect Dis. 2020 Oct;20(10):e274-e283. doi: 10.1016/S1473-3099(19)30742-X. Epub 2020 Jul 6. PMID 32645296
- [Derived] Madsen AMR, Gehrt L, Schaltz-Buchholzer F, Moller S, Christiansen R, Schellerup L, Norberg LA, Krause TG, Nielsen S, Bliddal M, Aaby P, Benn CS. Evaluating the effect of BCG vaccination for non-specific protection from infection in senior citizens during the COVID-19 pandemic: A randomised clinical trial. J Infect. 2024 Dec;89(6):106319. doi: 10.1016/j.jinf.2024.106319. Epub 2024 Oct 17. PMID 39423874

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from September 2020 to December 2021 in Odense, a Danish city of approximately 200,000 inhabitants. Citizens aged 65 years or older, with access to secure electronic mail from the authorities were eligible. Exclusion criteria were known contraindications to BCG vaccination.
Pre-assignment Details: Screening details:
  We screened 1,816 persons for inclusion; 140 fulfilled an exclusion criterion or declined to participate, and 1,676 were included and randomised to BCG (N=838) or placebo (N=838).
Groups:
- BCG-Denmark: Participants that are randomized to the active comparator arm will receive an adult 0.1 ml dose of BCG vaccine (BCG-Denmark, AJ Vaccines) in the skin covering the left upper deltoid muscle.
  Each 0.1 ml dose of vaccine contains between 200,000 to 800,000 colony forming units of the live attenuated strain of Mycobacterium bovis (BCG), Danish strain 1331.
  BCG-Denmark: Mycobacterium bovis BCG live attenuated BCG-Denmark vaccine (AJ Vaccines, Copenhagen, Denmark) administered by intradermal injection in the left deltoid region.
Period: Overall Study
Arm/Group | BCG-Denmark | Control
Started | 838 | 838
Completed | 838 | 838
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BCG-Denmark | Control | Total
Number analyzed (Participants) | 838 | 838 | 1676
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 838 | 838 | 1676
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70.5 [67.6 to 74.1] | 70.7 [67.9 to 74.1] | 70.6 [67.7 to 74.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 461 | 461 | 922
  Male | 377 | 377 | 754
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 838 | 838 | 1676
History of previous BCG vaccination [Count of Participants; unit: Participants] | 817 | 818 | 1635
Scar from previous BCG vaccination [Count of Participants; unit: Participants] | 717 | 725 | 1442
COVID-19 vaccinated before inclusion [Count of Participants; unit: Participants] — Received at least one dose of COVID-19 vaccine before enrolment.
  Participants | 180 | 174 | 354

OUTCOME MEASURES:

1. Primary Outcome: Acute Infection
Description: The primary outcome was a composite outcome of acute infection (recurrent events) defined as "infection attended by a physician", "use of antibiotics", "hospitalisation due to infection", or "death due to infection". All subcomponents were also analysed separately.
Time Frame: 12 months after inclusion
Measure: Number; unit: Events
Arm/Group | BCG-Denmark | Control
Number analyzed (Participants) | 838 | 838
Events
  Acute infection (composite) | 424 | 469
  Infection attended by a physician | 212 | 236
  Use of antibiotics | 338 | 341
  Hospitalisation due to infection | 23 | 29
  Death due to infection | 0 | 0
Statistical Analysis 1: Comparison: BCG-Denmark vs Control; Acute infection was analysed as recurrent events using an Andersen-Gill Cox proportional hazards regression model with time since inclusion as underlying time scale. The analysis was done for the composite outcome and for all subcomponents separately, presenting Hazard Ratios (HR) with 95% Confidence Intervals (CI) for each. For all recurrent outcomes, a wash-out period of 14 days was used to define new events; Test type: Superiority; p < 0.05, Andersen-Gill Cox

2. Secondary Outcome: Verified SARS-CoV-2 Infection (First Event)
Description: Verified SARS-CoV-2 infection was defined as having a positive SARS-CoV-2 Polymerase Chain Reaction (PCR) test or rapid antigen test.
Time Frame: 12 months after inclusion
Measure: Number; unit: Events
Arm/Group | BCG-Denmark | Control
Number analyzed (Participants) | 838 | 838
Events | 113 | 115
Statistical Analysis 1: Comparison: BCG-Denmark vs Control; Verified SARS-CoV-2 infection (first event) and all-cause hospitalisation (first event) was analysed using standard Cox proportional hazards models, but otherwise as described for primary outcome; Test type: Superiority; p < 0.05, Regression, Cox

3. Secondary Outcome: Self-reported Respiratory Symptoms (Recurrent Events)
Description: Self-reported respiratory symptoms were identified from questionnaires, where participants reported having had a respiratory illness such as common cold, influenza, pneumonia, or similar term, and/or reported one or more of the following symptoms: cough, sore throat, runny nose/nasal congestion (common cold symptoms), loss of smell or taste sense, or dyspnoea, with or without general symptoms such as fever, chills, muscle ache, headache, and fatigue (dyspnoea only if in combination with fever). This outcome also included symptoms not requiring medical attention.
Time Frame: 12 months after inclusion
Measure: Number; unit: Events
Arm/Group | BCG-Denmark | Control
Number analyzed (Participants) | 838 | 838
Events | 957 | 781
Statistical Analysis 1: Comparison: BCG-Denmark vs Control; The secondary outcome, self-reported respiratory symptoms, was analysed the same way as the primary outcome (recurrent events); Test type: Superiority; p < 0.05, Andersen-Gill Cox

4. Secondary Outcome: All-cause Hospitalisation (First Event)
Description: All-cause hospitalisation (first event) included all hospital admissions with overnight stay regardless of duration. Overnight stay was chosen as a condition to exclude contacts such as planned procedures and visits to outpatient clinics.
Time Frame: 12 months from inclusion.
Measure: Number; unit: Events
Arm/Group | BCG-Denmark | Control
Number analyzed (Participants) | 838 | 838
Events | 81 | 73
Statistical Analysis 1: Comparison: BCG-Denmark vs Control; Verified SARS-CoV-2 infection (first event) and all-cause hospitalisation (first event) was analysed using standard Cox proportional hazards models, but otherwise as described for the primary outcome; Test type: Superiority; p < 0.05, Regression, Cox

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events were registered within 14 days of randomisation. Serious adverse events until end of trial.
  Participants could report adverse events via the biweekly electronic questionnaires or directly to the investigators at all times during the trial.
Arm/Group | BCG-Denmark | Control
All-Cause Mortality (participants affected / at risk) | 1/838 | 3/838
Serious Adverse Events (participants affected / at risk) | 78/838 | 63/838
Other Adverse Events (participants affected / at risk) | 52/838 | 8/838
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCG-Denmark (N=838) | Control (N=838)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 8 (8)
Vascular (Vascular disorders) | 7 (7) | 7 (9)
Procedures (Surgical and medical procedures) | 0 (0) | 1 (1)
General disorders (General disorders) | 8 (8) | 8 (8)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Psichiatric disorders (Psychiatric disorders) | 1 (1) | 0 (0)
Injuries (Injury, poisoning and procedural complications) | 10 (10) | 3 (3)
Cardiac disorders (Cardiac disorders) | 19 (22) | 18 (20)
Neurological disorders (Nervous system disorders) | 0 (0) | 1 (1)
Eye disorders (Eye disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 8 (8) | 7 (9)
Hepatobiliary disorders (Hepatobiliary disorders) | 2 (2) | 0 (0)
Renal disorders (Renal and urinary disorders) | 2 (2) | 1 (1)
Musculoskeletal disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Infections (Infections and infestations) | 18 (20) | 11 (14)
Metabolic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCG-Denmark (N=838) | Control (N=838)
Vaccination site reactions (General disorders) | 52 (52) | 8 (8) — Local skin reactions and general reactions related to trial vaccination. Within 14 days of vaccination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT04542330/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT04542330/SAP_002.pdf